CLINICAL TRIAL: NCT00636883
Title: Oxaliplatin, Gemcitabine, and Erlotinib Study in Patients With Advanced Chemo-naïve Pancreatic Cancer
Acronym: GEMOX-T
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual rate
Sponsor: National Guard Health Affairs (Other Government)
Responsible Party: Principal Investigator, Nagham Sheblaq, CCRP, BsC. pharma, Senior Clinical Research Coordinator, King Abdulaziz Medical City
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC07/031
Record Dates: First submitted 2008-03-08; First posted 2008-03-17 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Oxaliplatin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gemcitabine — GEMOX-Erlotinib consists of erlotinib 100 mg orally daily starting day 1, Gemcitabine 1000 mg/m2 in 10 mg/m2/min (100 minutes) infusion on day 1 followed on day 2 by oxaliplatin 100 mg/m2 in a 2-hour infusion. Treatment will be repeated every 2 weeks. Each two weeks is a cycle.If at end of 12 cycles response continues, will administer Gemox and erlotinib till achieve maximum response. Then start Erlotinib maintenance therapy.
  Other Names: Oxaliplatin; Erlotinib

SUMMARY:
The purpose of this study is to determine if the combination of Gemcitabine, Oxaliplatin and Erlotinib in the treatment of patients with pancreatic cancer will provide increased clinical benefits and improvement in their quality of life.

DETAILED DESCRIPTION:
Treatment Plan GEMOX-Erlotinib consists of erlotinib 100 mg orally daily starting day 1, Gemcitabine 1000 mg/m2 in 10 mg/m2/min (100 minutes) infusion on day 1 followed on day 2 by oxaliplatin 100 mg/m2 in a 2-hour infusion. Treatment will be repeated every 2 weeks. Each two weeks is a cycle. Tumor response evaluation will be performed every 2 months. If tumor progress, patient will be off study, but if the disease is stable or PR, CR obtained will continue treatment for total of 12 cycles. If at end of 12 cycles response continues, will administer Gemox and erlotinib till achieve maximum response. Then start Erlotinib maintenance therapy.

Sample size: A total of 34 patients are needed assuming expected response is greater than 10% (about 27%) and a power = 80%. Fourteen patients will be treated in the first stage; if one patient achieved PR then additional twenty patients will be enrolled in the study for a total of 34 patients.

Statistical Methods: Response rate with 95% CI and median time to progression of disease will be calculated. Success will be declared if the lower limit of the 95% CI of the response rate is greater than 10%. The 95% CI of the response rate will be calculated using exact methods. Survival curve will be estimated using Kaplan-Meier Method. Descriptive statistics will be used to describe patient demographics, adverse events, serious adverse events and reasons for termination. Two approaches to the efficacy and safety analyses will be done; the ITT (intent-to-treat) for the efficacy analysis and safety. The ITT analysis consists of patients who received at least one dose of the study drug and at least one on-treatment measurement of the primary efficacy endpoint (overall response). The safety analysis consists of patients who received at least one dose of the study drug and at least one safety measurement done. A detailed description of the statistical methods, table and listing shells will be provided in the statistical analysis (SAP) before database lock or data transfer to the study biostatistician.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age between 18 and 75 years.
2. Presence of microscopic diagnosis of pancreatic cancer.
3. The disease is Locally advanced deemed by the surgeon to be unresectable, or metastatic disease.
4. Karnofsky Performance status >50%.
5. Prior radiotherapy for local diseases is allowed provided disease progression had been documented, and treatment completed at least 4 weeks before random assignment
6. Prior chemotherapy is not permitted, except for fluorouracil given concurrently as a radiosensitizer.
7. Patients must have normal organ function evidenced by

   * Cr <1.5 ULN
   * ANC >1000
   * platelets> 100,000
   * total bilirubin <1.5ULN.
8. Pain should be controlled for at least two weeks without an increase in the narcotic consumption.
9. Biliary obstruction should be controlled for at least two weeks evident by stable or improving liver function tests especially total bilirubin.
10. Patient has signed a Patient Informed Consent Form.
11. For all females of childbearing potential, a negative pregnancy test must be obtained within 72 hours before starting therapy.

Exclusion Criteria:

1. Contraindication to chemotherapy.
2. Evidence of uncontrolled CNS disease (patients with controlled CNS disease for 4 weeks using the same imaging method and for whom are off steroid will be eligible)
3. Uncontrolled Nausea and Vomiting
4. Diagnosis of other malignancy in the last 5 years excluding non-melanoma skin cancer and in -situ cervical cancer.
5. Subjects unlikely to comply with protocol, e.g. uncooperative attitude, inability to return for follow- up visits and unlikelihood of completing the study.
6. Any known history of hypersensitivity to the study drugs.
7. Pregnant or lactating women.
8. Participation in a clinical trial with any investigational drug used with curative intent and within 30 days prior to study entry
9. Peripheral sensitive neuropathy with functional impairment prior to study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Response rate (partial and complete response, stable disease, and progressive disease) | Tumor response will be assessed following the induction therapy and after cycle 4,8 and at the end of the treatment.

SECONDARY OUTCOMES:
Overall survival | UNMEASURABLE

CONTACTS AND LOCATIONS:
Overall Officials: Abdul-Rahman M Jazieh, MD,MPH, Principal Investigator — National Guard Hospital Affairs
Locations (1):
- National Guard Health Affairs, Riyadh, Saudi Arabia